CLINICAL TRIAL: NCT00639353
Title: The Clinical Performance of the Silicone Hydrogel Contact Lens on Low to Moderate Astigmatism in Japan
Brief Title: Silicone Hydrogel Contact Lenses on Low Astigmatism in Japan
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: English to Japanese translation issues caused enrollment of incorrect and unqualified subjects; error applied to all subjects enrolled prior to termination.
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-0804
Record Dates: First submitted 2008-03-14; First posted 2008-03-20 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Refractive Error; Myopia; Astigmatism
MeSH Terms: conditions — Refractive Errors; Myopia; Astigmatism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- spherical contact lens (Active Comparator): Subjects will wear and evaluate a spherical soft contact lens daily for 2 weeks
  Interventions: Device: senofilcon A sphere soft contact lens
- toric contact lens (Experimental): Subjects will wear and evaluate a toric soft contact lens daily for 2 weeks
  Interventions: Device: senofilcon A toric soft contact lens

INTERVENTIONS:
Device: senofilcon A toric soft contact lens — contact lens
  Other Names: ACUVUE OASYS for Astigmatism
  Arms: toric contact lens
Device: senofilcon A sphere soft contact lens — contact lens
  Other Names: ACUVUE OASYS
  Arms: spherical contact lens

SUMMARY:
This study seeks to evaluate the clinical performance of a recently released contact lens designed to correct astigmatism to an established contact lens that has historically been used in these patients.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is 18 to 39 years of age. (Parental consent is required for a minor child i.e. under the age of 20.)
2. The subject has signed an informed consent with his/her own judgement for participation in the study.
3. The subject currently is a habitual wearer of spherical or toric daily-wear soft contact lenses, excluding daily disposables, in daily wear bases.

Exclusion Criteria:

1. The subject has any ocular or systemic allergies that interfere with contact lens wear.
2. The subject has dry eye and lacrimal apparatus disease that could interfere with contact lens wear.
3. The subject has any systemic disease or autoimmune disease that interferes with contact lens wear.
4. The subject has corneal edema, neovascularization, corneal staining or other ocular abnormalities (Grade 3 or above) that clinically apparently interfere with contact lens wear.
5. The subject has any anterior segment eye disease (palpebral abnormalities, corneal hypesthesia, corneal epithelial defect, bulbar conjunctival hyperemia, etc.) that clinically apparently interferes with contact lens wear.
6. The subject has a history of solution reactions to the chemical cleaner/disinfectant to be used in this study, as far as known to the subject.
7. The subject has ocular infection.
8. The subject has ocular inflammation (including acute/subacute anterior segment inflammations and uveitis).
9. The subject has corneal distortion resulting from previous experience of hard contact lens wear.
10. The subject has infectious disease (pneumonia, tuberculosis, etc.) or immunosuppressive disease (HIV positive etc.), as far as known to the subject.
11. The subject has diabetes, as far as known to the subject.
12. The subject is pregnant or in the lactation period, as far as known to the subject.
13. The subject uses any eye remedies (excluding artificial tear substitutes or hyaluronic acid drops for reducing dryness while wearing contact lenses).
14. The subject had any ocular trauma or surgery within 8 weeks prior to participation in the study.
15. The subject is a wearer of hard contact lenses (including rigid gas permeable).
16. The subject is exposed to a dry environment on a constant basis.
17. The subject is exposed to a living environment where dust, chemicals, etc. can easily enter the eye.
18. The subject is unable to follow the principal investigator's instructions.
19. The subject is unable to follow lens hygiene procedures necessary for contact lens wear.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2008-02; Primary Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Subject-reported satisfaction for vision | After 2 weeks of lens wear
  Scale of 0 to 100, were 0=extremely poor and 100=Excellent
Subject-reported satisfaction for comfort. | After 2 weeks of lens wear
  Scale of 0 to 100, were 0=extremely poor and 100=Excellent

SECONDARY OUTCOMES:
Subject preference for lens type. | After 2 weeks of lens wear.

CONTACTS AND LOCATIONS:
Locations (10):
- Japan (10):
  - Shioya eye clinic, Fukushima, Fukushima
  - Takahashi eye clinic, Odawarashi, Kanagawa
  - Kodama eye clinic, Jyoyoshi, Kyoto
  - Inaba eye clinic, Osakashi, Osaka
  - Iwasaki eye clinic, Osakashi, Osaka
  - Watanabe eye clinic, Osakashi, Osaka
  - Sakura eye clinic, Shizuoka, Shizuoka
  - Kajita eye clinic, Minatoku, Tokyo
  - Dogenzakaitoi eye clinic, Shibuyaku, Tokyo
  - Ueda eye clinic, Shimonosekishi, Yamaguchi